CLINICAL TRIAL: NCT02494089
Title: Analysis of the Stress Induced by in Situ Simulation
Acronym: SIMSTRESS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Principal Investigator, Yannick BRUNIN, Doctor, Centre Hospitalier Universitaire de Besancon
Other Study IDs: SIM STRESS
Record Dates: First submitted 2015-05-29; First posted 2015-07-10 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Psychologic Stress; Heart Arrest
Keywords: in situ simulation; in hospital cardiac arrest; clinical audit; education; patient simulation
MeSH Terms: conditions — Stress, Psychological; Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: distress analysis

SUMMARY:
Vulnerability to psychologic distress induced by in situ simulation.

Objectives: Psychological evaluation at short and long term on working satisfaction, mental health, and acute stress after in situ simulation. Analysis of the stress vulnerability induced by simulation.

Design: non interventional study.

Primary outcome: Psychologic distress analysis with validated psychologic distress inventory (Job Satisfaction Survey (JSS), General Health Quality (GHQ), Impact of Event Scale Revisited (IESR), State-Trait Anxiety Inventory-A (STAI-A), State-Trait Anxiety Inventory -B (STAI-B)).

ELIGIBILITY:
Inclusion Criteria:

* team members: nurses, auxiliary nurse, residents, doctors, students

Exclusion Criteria:

* non volunteers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: team members
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
psychologic distress analysis induced by in situ simulation | 3 weeks
  auto-validated distress inventory: IESR-R STAI-A STAI-B GHQ-12 JSS

SECONDARY OUTCOMES:
Stress vulnerability to in situ simulation | 3 weeks
  distress inventory: JSS STAI-A social questionary